CLINICAL TRIAL: NCT00447590
Title: Effectiveness and Safety Study of LAP-BAND Treatment for Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBA-001
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

ARMS (1):
- LAP-BAND (Experimental): All subjects who received the LAP-BAND System.
  Interventions: Device: LAP-BAND System

INTERVENTIONS:
Device: LAP-BAND System — Restriction of food intake

SUMMARY:
The purpose of this study is to determine whether the LAP-BAND system is safe and effective in morbidly obese adolescents.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety and effectiveness of the LAP-BAND System in a morbidly obese adolescent population, ages 14 to 17 years. The secondary objectives were to assess associated changes from baseline in obesity-related comorbidities as well as psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14 and 17 at the time of enrollment
* Have a BMI ≥ 40 kg/m2 (with or without obesity-related co-morbid conditions) or BMI ≥ 35 kg/m2 with one or more severe co-morbid conditions
* Have a history of obesity for at least 2 years and have failed more conservative weight-reduction alternatives, such as supervised diet, exercise and behavior modification programs

Exclusion Criteria:

* Family or subject history of congenital or acquired anomalies of the gastrointestinal tract
* Severe cardiopulmonary or other serious or uncontrolled organic disease
* Severe coagulopathy; hepatic insufficiency or cirrhosis
* History of bariatric, gastric, or esophageal surgery
* History of intestinal obstruction or adhesive peritonitis
* History of esophageal dysmotility disorders
* Type I diabetes

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apollo Endosurgery, Study Director — Apollo Endosurgery, Inc.
Locations (1):
- Apollo Endosurgery, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 174 participants were enrolled in the study, where enrollment was defined as signing the informed consent form.
  21 participants were not implanted after signing the informed consent. 153 participants were treated with the LAP-BAND.
Period: Overall Study
Arm/Group | LAP-BAND
Started | 153 (153 participants were treated with the LAP-BAND System.)
Completed | 93 (Completing the study was defined as the number of participants in the study at month 60 (5 years).)
Not Completed | 60
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 24
Not completed — Band Removed/Eroded/Other Follow-Up Loss | 10

BASELINE CHARACTERISTICS:
Population: The baseline population consisted of all subjects who were implanted with the LAP-BAND System.
Arm/Group | LAP-BAND
Number analyzed (Participants) | 153
Age, Continuous [Mean (Full Range); unit: years] | 15.8 [14 to 18]
Age, Customized [Number; unit: participants]
  Age 14 | 25
  Age 15 | 33
  Age 16 | 47
  Age 17 | 46
  Age 18 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 102
  Black/African-American | 37
  Hispanic/Latino | 10
  Other | 4
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m2] | 48.5 [34.0 to 73.3]
Excess Weight [Mean (Full Range); unit: pounds (lb)] — Excess weight is equal to operative weight minus ideal weight at visit.
  pounds (lb) | 152.3 [51.8 to 346.9]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Attain Clinically Successful Weight Loss of ≥30% Excess Weight Loss (EWL) at 1 Year Post LAP-BAND Implantation.
Description: Percent Excess Weight Loss was defined as Weight Loss divided by Excess Weight multiplied by 100.
  Excess Weight = baseline weight - ideal weight, where Ideal weight was determined using the 85th percentile on the Centers for Disease Control (CDC) Growth Charts for children and adolescents ages 2 to 20 years.
Time Frame: 1 year
Population: Intent to treat (ITT) population with imputation at month 12 (ITT population consisted of participants treated with the LAP-BAND).
Measure: Number; unit: percentage of participants
Arm/Group | LAP-BAND
Number analyzed (Participants) | 153
percentage of participants | 49.7
Statistical Analysis 1: Comparison: LAP-BAND; p-Value is from a 2-sided exact binomial test to test the null hypothesis that 30% of subjects have at least 30% EWL; Test type: Superiority or Other; p < 0.0001, 2-sided Exact Binomial Test

2. Secondary Outcome: Subject Excess Weight Loss Throughout the Study
Description: Excess Weight Loss was examined over the 5 year period post LAP-BAND implantation. Excess Weight Loss was defined as Weight Loss divided by Excess Weight multiplied by 100.
Time Frame: Baseline to 5 Years
Population: Intent to treat (ITT) population with imputation at month 60
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | LAP-BAND
Number analyzed (Participants) | 153
%EWL | 27.0 (45.46) [19.69 to 34.21]

3. Secondary Outcome: Subject Percent Excess BMI Loss
Description: Subject Percent Excess BMI Loss was examined at 5 years post LAP-BAND placement.
Time Frame: Baseline to 5 Years
Population: Intent to treat (ITT) population with imputation at month 60
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | LAP-BAND
Number analyzed (Participants) | 153
kg/m2 | -6.0 (11.12) [-7.41 to -4.62]

4. Secondary Outcome: Change in Subjects' Comorbid Conditions
Description: The change from baseline to year five in subjects' comorbid conditions of Type II Diabetes, Dyslipidemia, and Hypertension. Change as reported below indicates the condition resolved.
Time Frame: Baseline to 5 Years
Population: Subjects who had a specific comorbid condition at baseline (Diabetes n=9, Dyslipidemia n=39, Hypertension n=22)
Measure: Number; unit: participants whose condition resolved
Arm/Group | LAP-BAND
Number analyzed (Participants) | 70
participants whose condition resolved
  Diabetes Type II (n=9) | 3
  Dyslipidemia (n=39) | 14
  Hypertension (n=22) | 7

5. Secondary Outcome: Change in Quality of Life Using the Beck Depression Inventory II (BDI)
Description: Quality of life was examined using the Beck Depression Inventory II (BDI) questionnaire, which scores on a range from 0 (best) to 63 (worst). The change in subjects' BDI II score was assessed from baseline to 5 years.
Time Frame: Baseline to 5 Years
Population: Participants who completed the BDI II questionnaire through month 60
Measure: Mean (95% Confidence Interval); unit: units on BDI scale
Arm/Group | LAP-BAND
Number analyzed (Participants) | 74
units on BDI scale | -1.0 [-2.64 to 0.39]

6. Secondary Outcome: Change in Quality of Life Using Impact of Weight on Quality of Life (IWQOL) Kids Questionnaire
Description: Quality of life was examined using the Impact of Weight on Quality of Life (IWQOL) Kids questionnaire, which has a score range from 0(worst) to 100(best). The change in subjects' IWQOL Kids score was assessed from baseline to 5 years.
Time Frame: Baseline to 5 Years
Population: Participants who completed the IWQOL Kids questionnaire through month 60 (year 5).
Measure: Mean (95% Confidence Interval); unit: units on IWQOL Kids scale
Arm/Group | LAP-BAND
Number analyzed (Participants) | 72
units on IWQOL Kids scale | 18.0 [14.42 to 21.59]

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected from the time of LAP-BAND implantation to 5 years (end of study).
Description: Device-related Serious Adverse Events (SAEs) and Adverse Events (AEs) are reported. AEs occurring with frequency of >=1% are reported.
Arm/Group | LAP-BAND
Serious Adverse Events (participants affected / at risk) | 20/153
Other Adverse Events (participants affected / at risk) | 133/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND (N=153)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Band Slip (Gastrointestinal disorders) | 9 (9)
Band erosion (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Esophageal irritation (Gastrointestinal disorders) | 1 (1)
Esophagus distended (Gastrointestinal disorders) | 1 (1)
Gastric erosion (Gastrointestinal disorders) | 1 (1)
Gastric herniation via Lap-Band (Gastrointestinal disorders) | 1 (1)
Gastric prolapse (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 2 (2)
Intra-abdominal sepsis (Gastrointestinal disorders) | 1 (2)
Large gastric pouch (Gastrointestinal disorders) | 1 (1)
Port Tubing disconnect (Surgical and medical procedures) | 2 (2)
Possible acute obstruction of the Lap-Band (Gastrointestinal disorders) | 1 (1)
Recurrent pouch enlargement (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Surgical site infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND (N=153)
Vomiting (Gastrointestinal disorders) | 83 (83)
Gastric dilatation (Gastrointestinal disorders) | 62 (62)
Dysphagia (Gastrointestinal disorders) | 38 (38)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 31 (31)
Abdominal pain (Gastrointestinal disorders) | 30 (30)
Nausea (Gastrointestinal disorders) | 30 (30)
Dyspepsia (Gastrointestinal disorders) | 28 (28)
Oesophageal dilatation (Gastrointestinal disorders) | 26 (26)
Abdominal pain upper (Gastrointestinal disorders) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 12 (12)
Hiatus hernia (Gastrointestinal disorders) | 8 (8)
Medical device complication (Injury, poisoning and procedural complications) | 24 (24)
Post procedural pain (Injury, poisoning and procedural complications) | 14 (14)
Device failure (Injury, poisoning and procedural complications) | 12 (12)
Implant site pain (General disorders) | 8 (8)
Non-cardiac chest pain (General disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No